CLINICAL TRIAL: NCT03439007
Title: Prediction of Hypotension During Induction of Anesthesia in Pediatric Patients Using Dynamic Variables of Fluid Responsiveness
Brief Title: Anesthesia-induced Hypotension and Fluid Responsiveness
Acronym: PVI
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Prof., Seoul National University Hospital
Other Study IDs: 1712-091-907
Record Dates: First submitted 2018-01-27; First posted 2018-02-20 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Hypotension on Induction
Keywords: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotensive: A group of pediatric patients who showed hypotension during induction of anesthesia
- Normotensive: A group of pediatric patients who did not show hypotension during induction of anesthesia

SUMMARY:
The purpose of this study is to find out which of the variables related to fluid responsiveness (e. g., perfusion index [PI], pleth variability index [PVI], pulse oximetry plethysmographic variance [ΔPOP]) can best predict hypotension during induction of anesthesia.

DETAILED DESCRIPTION:
Propofol is a widely used intravenous agent for induction of anesthesia in children aged 3 years and more. A well-known adverse effect of propofol is hypotension, which can be properly dealt with hydration and/or administration of inotropics and vasopressors. However, severe hypotension during anesthetic induction may not be immediately cured if anesthesiologist should concentrate on ventilation of the patient. Since pediatric patients have smaller reservoir for oxygen supply and perfusion to various organs of the body, delayed handling of severe hypotension may result in irreversible damage to the vital organs.

Hypotension during anesthesia is caused, though not entirely, by dehydration. There are a variety of non-invasive variables that are related to the severity of dehydration, but which of the variables can best predict anesthesia-induced hypotension in pediatric patients. In this study, we will measure the preoperative values of non-invasive variables related to fluid status, and find out which of them are most closely related to the occurrence of hypotension during anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-6 years
* Scheduled to undergo elective surgery under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification III or more
* Contraindication of laryngeal mask airway (LMA) insertion:

  (1) Esophagitis, gastritis, peptic ulcer, pyloric or intestinal stenosis, history of upper gastrointestinal tract surgery, body mass index [BMI] > 30, expected anesthesia time > 2 hours)
* Arrhythmia
* Left ventricular failure (ejection fraction < 40%)
* Congenital syndromes which are known to affect cardiopulmonary function
* Use of inotropics/vasopressors before anesthesia
* History of allergic reaction to drugs used in general anesthesia

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3-6 years
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pleth variability index | changes for 10 minutes
  pleth variability index

SECONDARY OUTCOMES:
Adverse event_1 | 10 minutes
  bradycardia
Adverse event_2 | 10 minutes
  hypotention
Adverse event_3 | 10 minutes
  EEG changes
Adverse event_4 | 10 minutes
  desaturation < 95%
Heart rate | changes for 10 minutes
  heart rate
perfusion index | changes for 10 minutes
  perfusion index
pulse oximetry plethysmograpic variance | changes for 10 minutes
  pulse oximetry plethysmograpic variance

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided